CLINICAL TRIAL: NCT01528787
Title: A Phase 2, Double-masked, Randomized, Placebo-controlled, Dose-response Study Assessing the Safety and Ocular Hypotensive Efficacy of Three Doses of AR-13324 Ophthalmic Solution in Patients With Elevated Intraocular Pressure
Brief Title: Study of AR-13324 in Patients With Elevated Intraocular Pressure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aerie Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AR-13324-CS201
Record Dates: First submitted 2012-02-05; First posted 2012-02-08 (Estimated); Results first posted 2018-02-22 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2016-06

CONDITIONS: Ocular Hypertension; Open Angle Glaucoma
Keywords: Intraocular pressure; visual field; Ocular hypertension or open angle glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle | interventions — netarsudil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- AR-13324 Ophthalmic Solution 0.01% (Experimental): 1 drop to study eye once daily
  Interventions: Drug: AR-13324 Ophthalmic Solution 0.01%
- AR-13324 Ophthalmic Solution 0.02% (Experimental): 1 drop to study eye once daily
  Interventions: Drug: AR-13324 Ophthalmic Solution 0.02%
- AR-13324 Ophthalmic Solution 0.04% (Experimental): 1 drop to study eye once daily
  Interventions: Drug: AR-13324 Ophthalmic Solution 0.04%
- AR-13324 Ophthalmic Solution Vehicle (Placebo Comparator): 1 drop to study eye once daily
  Interventions: Other: AR-13324 Ophthalmic Solution Vehicle

INTERVENTIONS:
Drug: AR-13324 Ophthalmic Solution 0.01% — Administered to study eye, once daily (QD) in the morning (AM) for 7 days
  Arms: AR-13324 Ophthalmic Solution 0.01%
Drug: AR-13324 Ophthalmic Solution 0.02% — Administered to study eye, QD AM for 7 days
  Other Names: Netarsudil
  Arms: AR-13324 Ophthalmic Solution 0.02%
Drug: AR-13324 Ophthalmic Solution 0.04% — Administered to study eye, QD AM for 7 days
  Arms: AR-13324 Ophthalmic Solution 0.04%
Other: AR-13324 Ophthalmic Solution Vehicle — Administered to study eye, QD AM for 7 days
  Arms: AR-13324 Ophthalmic Solution Vehicle

SUMMARY:
In this double-masked, vehicle-controlled, dose-response study, subjects will be randomized to receive AR-13324 Ophthalmic Solution 0.01%, 0.02%, and 0.04% or its vehicle (one eye), once daily (QD)in the morning (AM) for 7 days. The first dose and last dose will be administered in the clinic. Ocular safety and ocular hypotensive efficacy will be evaluated in the clinic throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or greater. 18 years of age or greater.
2. Diagnosis of open angle glaucoma (OAG) or ocular hypertension (OHT).
3. Unmedicated (post-washout, p.r.n.) IOP ≥ 24 mm Hg in one or both eyes at 08:00 hours, ≥ 21 mm Hg at 10:00, 12:00 and 16:00 hours on post-washout measurement (Visit 1).
4. Corrected visual acuity in each eye +1.0 logMAR or better by ETDRS in each eye (equivalent to 20/200).
5. Able and willing to give signed informed consent and follow study instructions.

Exclusion Criteria:

Ophthalmic: Either eye

1. Intraocular pressure > 36 mm Hg
2. Known hypersensitivity to any component of the formulation or to topical anesthetics, (benzalkonium chloride, etc.)
3. Ocular trauma within the past six months, or ocular surgery or laser treatment within the past three months.
4. Evidence of ocular infection, inflammation, clinically significant blepharitis or conjunctivitis at baseline (Visit 1), or history of herpes simplex keratitis.
5. Contact lens wear within 30 minutes of instillation of study medication.
6. Ocular medication of any kind within 30 days of Visit 2, with the exception of a) ocular hypotensive medications (which must be washed out according to the provided schedule), b) lid scrubs (which may be used prior to, but not after Visit 2) or c) lubricating drops for dry eye (which may be used throughout the study),
7. Clinically significant ocular disease (e.g. corneal edema, uveitis, severe keratoconjunctivitis sicca) which might interfere with the study, including glaucomatous damage so severe that washout of ocular hypotensive medications for one month is not judged safe (e.g., advanced glaucomatous optic nerve head or visual field loss).
8. Any abnormality preventing reliable applanation tonometry in either eye. Study eye:
9. Glaucoma: pseudoexfoliation or pigment dispersion component, history of acute angle-closure glaucoma, or closed or narrow angle upon gonioscopy. Note: Previous laser peripheral iridotomy is NOT acceptable.
10. Previous glaucoma intraocular surgery or laser procedures such as argon laser trabeculoplasty (ALT), selective laser trabeculoplasty (SLT) or micropulse laser trabeculoplasty ( MLT), as well as refractive procedures such as radio keratotomy (RK), laser eye surgery (LASIK), photorefractive keratectomy (PRK), or collagen cross linking.
11. Central corneal thickness greater than 600 μm.

    General/Systemic:
12. Clinically significant abnormalities in laboratory tests at screening, recognizing that subjects are not fasting at the time of drawing blood.
13. Clinically significant systemic disease (e.g., uncontrolled diabetes, myasthenia gravis, hepatic, renal, cardiovascular or endocrine disorders) which might interfere with the study.
14. Participation in any investigational study within the past 30 days.
15. Changes of systemic medication during the study that could have a substantial effect on IOP within 30 days prior to screening, or anticipated during the study.
16. Due to status of preclinical safety program, women of childbearing potential who are pregnant, nursing, planning a pregnancy, or not using a medically acceptable form of birth control. An adult woman is considered to be of childbearing potential unless she is one year post-menopausal or three months post-surgical sterilization. All females of childbearing potential must have a negative urine pregnancy test result at the screening examination and must not intend to become pregnant during the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2012-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Heah, MD, Study Director — Aerie Pharmaceuticals, Inc.
Locations (11):
- United States (11):
  - Aesthetic Eye Care Institute, Newport Beach, California
  - Robert Noecker, M.D., M.B.A., Fairfield, Connecticut
  - Coastal Research Associates, LLC, Roswell, Georgia
  - Heart of America Eye Care, P.A., Shawnee Mission, Kansas
  - Comprehensive Eye Care, St Louis, Missouri
  - Rochester Ophthalmology Group, Rochester, New York
  - The Eye Institute, Tulsa, Oklahoma
  - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Univ Eye Surgeons, Maryville Ctr., Maryville, Tennessee
  - Texan Eye, Austin, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- AR-13324 Ophthalmic Solution 0.01%; AR-13324 Ophthalmic Solution 0.02%; AR-13324 Ophthalmic Solution 0.04%; AR-13324 Opththalmic Solution Vehicle: 1 drop to study eye once daily (QD) in the morning (AM)
Period: Overall Study
Arm/Group | AR-13324 Ophthalmic Solution 0.01% | AR-13324 Ophthalmic Solution 0.02% | AR-13324 Ophthalmic Solution 0.04% | AR-13324 Opththalmic Solution Vehicle
Started | 22 | 21 | 19 | 23
Completed | 22 | 21 | 18 | 22
Not Completed | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Family Emergency | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- AR-13324 Ophthalmic Solution Vehicle: 1 drop to study eye once daily (QD) in the morning (AM)
- Total: Total of all reporting groups
Arm/Group | AR-13324 Ophthalmic Solution 0.01% | AR-13324 Ophthalmic Solution 0.02% | AR-13324 Ophthalmic Solution 0.04% | AR-13324 Ophthalmic Solution Vehicle | Total
Number analyzed (Participants) | 22 | 21 | 19 | 23 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (12.36) | 69.1 (8.69) | 66.1 (11.09) | 57.8 (12.27) | 64.0 (11.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 10 | 13 | 51
  Male | 8 | 7 | 9 | 10 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 2 | 4 | 11
  Not Hispanic or Latino | 18 | 20 | 17 | 19 | 74
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 2 | 2 | 8
  White | 20 | 17 | 17 | 20 | 74
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP)
Description: The primary efficacy outcome was the mean IOP across subjects within treatment group at each post-treatment timepoint of Day 8.
  Instillation of study treatment commenced on Day 2 following measurement of IOP. IOP was measured at 0800, 1000, 1200 and 1600 hours on days 2 and 8. IOP was also measured at 0800 hours on Day 4.
Time Frame: Study treatment was administered for 7 days; starting on Day 2 and ending on Day 8.
Population: Modified intent to treat (mITT) population (85 patients receiving investigational treatment). Participants who did not complete the study did not contribute data at later time points.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AR-13324 Ophthalmic Solution 0.01% | AR-13324 Ophthalmic Solution 0.02% | AR-13324 Ophthalmic Solution 0.04% | AR-13324 Ophthalmic Solution Vehicle
Number analyzed (Participants) | 22 | 21 | 19 | 23
mmHg
  Day 2, 0800 hours | 25.80 (3.699) | 26.02 (2.542) | 26.50 (3.358) | 25.17 (2.980)
  Day 2, 1000 hours | 22.45 (3.713) | 22.10 (3.149) | 24.29 (5.347) | 22.87 (2.681)
  Day 2, 1200 hours | 21.93 (2.997) | 21.95 (3.653) | 25.00 (5.292) | 22.91 (2.863)
  Day 2, 1600 hours | 20.70 (3.521) | 20.88 (3.467) | 22.29 (4.849) | 21.41 (3.110)
  Day 4, 0800 hours: number analyzed (Participants) | 22 | 21 | 19 | 22
  Day 4, 0800 hours | 21.32 (4.049) | 21.00 (4.530) | 22.00 (5.352) | 23.98 (3.730)
  Day 8, 0800 hours: number analyzed (Participants) | 22 | 21 | 18 | 22
  Day 8, 0800 hours | 20.82 (5.487) | 20.60 (3.491) | 20.44 (3.933) | 24.34 (3.663)
  Day 8, 1000 hours: number analyzed (Participants) | 22 | 21 | 18 | 22
  Day 8, 1000 hours | 18.20 (4.165) | 18.71 (3.208) | 19.42 (3.663) | 22.34 (4.034)
  Day 8, 1200 hours: number analyzed (Participants) | 22 | 21 | 18 | 22
  Day 8, 1200 hours | 17.57 (4.255) | 17.88 (3.457) | 18.78 (4.486) | 21.93 (3.818)
  Day 8, 1600 hours: number analyzed (Participants) | 22 | 21 | 18 | 22
  Day 8, 1600 hours | 17.68 (3.161) | 16.88 (3.049) | 17.83 (3.510) | 21.52 (4.244)

ADVERSE EVENTS:
Arm/Group | AR-13324 Ophthalmic Solution 0.01% | AR-13324 Ophthalmic Solution 0.02% | AR-13324 Ophthalmic Solution 0.04% | AR-13324 Ophthalmic Solution Vehicle
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/21 | 0/19 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21 | 0/19 | 0/23
Other Adverse Events (participants affected / at risk) | 12/22 | 15/21 | 17/19 | 1/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AR-13324 Ophthalmic Solution 0.01% (N=22) | AR-13324 Ophthalmic Solution 0.02% (N=21) | AR-13324 Ophthalmic Solution 0.04% (N=19) | AR-13324 Ophthalmic Solution Vehicle (N=23)
Conjunctival Hyperaemia (Eye disorders) | 11 | 12 | 14 | 1
Ocular Hyperaemia (Eye disorders) | 1 | 1 | 3 | 0
Erythema of Eyelid (Eye disorders) | 0 | 1 | 1 | 0
Vision Blurred (Eye disorders) | 0 | 2 | 1 | 0
Diplopia (Eye disorders) | 0 | 0 | 1 | 0
Dry Eye (Eye disorders) | 0 | 2 | 0 | 0
Vitreous Floaters (Eye disorders) | 0 | 0 | 1 | 0
Instillation Site Reaction (General disorders) | 0 | 0 | 2 | 0
Corneal Staining (Investigations) | 0 | 2 | 1 | 0
Blood Glucose Increased (Investigations) | 0 | 1 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No